CLINICAL TRIAL: NCT06147622
Title: A Phase 1, Open-label, Cross-over Study in Healthy Volunteers to Assess the Pharmacokinetic Profile of Prazosin and Cyproheptadine Following Single Dose Oral Administration of KT110 Tablet and Following Administration of Alpress and Periactin Marketed Tablets
Brief Title: A Study to Assess the Pharmacokinetic Profile of Prazosin and Cyproheptadine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinnov Therapeutics (Other)
Responsible Party: Sponsor
Organization: Greenpharma S.A.S. (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OP111821.KIN
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Prazosin; Cyproheptadine

STUDY DESIGN:
Intervention Model Description: open-label, randomized, 2-period, single dose, crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT110 (Experimental): Subjects will be randomized to receive KT110 on period 1 or period 2
  Interventions: Drug: KT110
- Prazosin + cyproheptadine (Experimental): Subjects will be randomized to receive prazosin + cyproheptadine on period 1 or period 2
  Interventions: Drug: Prazosin + cyproheptadine

INTERVENTIONS:
Drug: Prazosin + cyproheptadine — Subjects will receive prazosin + cyproheptadine on day 1 of period 1 or on day 1 of period 2 depending on randomization.
  Arms: Prazosin + cyproheptadine
Drug: KT110 — Subjects will receive KT110 on day 1 of period 1 or on day 1 of period 2 depending on randomization.
  Arms: KT110

SUMMARY:
The study is an open-label, randomized,2-period, single dose, crossover study in 8 healthy male/female volunteers. Subjects will be randomized to the following sequences:

(A) Period 1: KT110 - wash-out period - Period 2: Alpress and Periactin marketed tablets ; Or (B) Period 1: Alpress and Periactin marketed tablets - wash-out period - Period 2: KT110

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female subject
* Females of childbearing potential and male participant must agree to use an adequate and highly effective method of contraception
* Negative serum pregnancy test at screening for woman of childbearing potential only
* Non-smoker subject or smoker of not more than 5 cigarettes a day
* Body Mass Index (BMI) between 18.5 and 30 kg/m2 inclusive, at screening

Exclusion Criteria:

* Any contraindication to Prazosin or Cyproheptadine treatments;
* Frequent headaches and / or migraine, recurrent nausea and / or vomiting;
* Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease equal to or greater than 20 mmHg in systolic blood pressure (SBP) and a decrease equal to or greater than 10 mmHg in diastolic blood pressure (DBP) within two minutes of changing from supine to standing position;
* Blood donation (including as part of a clinical trial) in the 2 months before administration
* Any drug intake (except paracetamol or contraception) during the month prior to the first administration;
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day)
* Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day);
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C Virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
* Positive results of screening for drugs of abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) 0-t | Day 4
  Area under the curve from time 0 to the last measurable concentration at time t
AUC 0-inf | Day 4
  Area under the curve from time 0 extrapolated to infinity (only for Cyproheptadine)
Cmax | Day 4
  Maximum observed concentration
Tmax | Day 4
  Time of maximum observed concentration
T1/2 | Day 4
  Apparent elimination half-life
K el | Day 4
  Apparent Elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No